CLINICAL TRIAL: NCT02032056
Title: The Effect of Probiotics in Reducing Infections and Allergic Manifestations in Young Children During the Complementary Feeding Period
Brief Title: Effect of Probiotics in Reducing Infections and Allergies in Young Children During the Complementary Feeding Period
Acronym: ProbiComp
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Changes in study design
Sponsor: University of Copenhagen (Other)
Collaborators: The Danish Council for Strategic Research (Other); Chr Hansen (Industry); Technical University of Denmark (Other); University of Bergen (Other); Odense University Hospital (Other); Statens Serum Institut (Other)
Responsible Party: Principal Investigator, Arne Astrup, Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-3-2013-064; H-3-2013-064 (Other Grant/Funding Number: The Danish Council for Strategic Research)
Record Dates: First submitted 2013-11-20; First posted 2014-01-09 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Days Absent From Day Care; Respiratory Tract Infections; Gastrointestinal Infections; Allergy
Keywords: Infections; Allergy; Immune function; Microbiota; infant
MeSH Terms: conditions — Respiratory Tract Infections; Hypersensitivity; Infections | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- probiotic (10^9 cfu/day) (Experimental): Daily intake of bifidobacterium animalis ssp. Lactis (BB12), 10^9 cfu/day, provided as powder in a sachet which can be added to food or drink.
  Interventions: Dietary Supplement: Probiotic (10^9 CFU/day)
- probiotic (10^8 cfu/day) (Experimental): Daily intake of bifidobacterium animalis ssp. Lactis (BB12), 10^8 cfu/day, provided as powder in a sachet which can be added to food or drink.
  Interventions: Dietary Supplement: Probiotic (10^8 CFU/day)
- Placebo (Placebo Comparator): provided as powder in a sachet which can be added to food or drink.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic (10^9 CFU/day)
  Other Names: Bifidobacterium animalis ssp. Lactis (BB12)
  Arms: probiotic (10^9 cfu/day)
Dietary Supplement: Probiotic (10^8 CFU/day)
  Other Names: Bifidobacterium animalis ssp. Lactis (BB12)
  Arms: probiotic (10^8 cfu/day)
Other: Placebo
  Arms: Placebo

SUMMARY:
The aim of the intervention is to examine the effect of the bacterial strain BB-12, provided for 6 mo, on the prevalence of infections and allergic manifestations in small children, and how BB-12 affects the immune system, the gastrointestinal tract and the microbiota. Children are enrolled during 2 winter seasons.

ELIGIBILITY:
Inclusion Criteria:

* 9 - 12 1/2 month at intervention start
* Start in daycare 4 +/- 2 weeks after intervention start
* Single born

Exclusion Criteria:

* Children born before 37th gestational week
* Children with a birth weight < 2500 g
* Children suffering from severe chronic illness
* Children receiving regular medication
* Children who have received antibiotics within a month before intervention start
* Children whose parents do not speak Danish

Ages: 9 Months to 13 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of days absent from day care due to respiratory and gastrointestinal infections | Up to 6 month
  Recorded weekly by the parents using web-based questionnaires

SECONDARY OUTCOMES:
Acute upper respiratory tract infections | Up to 6 month
  Number of days with acute upper respiratory tract infections (URTI); Number of children with at least 1 episode of URTI; Number of children with at least 3 episodes of URTI; Number of URTI episodes/child/year; Duration of URTI episodes (days);
  Additionally,symptoms of cold (defined as 2 days with runny/stuffy nose or cough)
  Recorded by the parents daily/weekly using web-based questionnaires.
Acute lower respiratory infections | Up to 6 month
  Number of children with at least 1 episode of a lower respiratory tract infection (LRTI).
  LRTI include bronchitis and pneumonia
  Recorded by the parents weekly using web-based questionnaires.
Gastrointestinal infections | Up to 6 month
  Number of children with at least 1 episode of diarrhea; Duration of episodes with diarrhea(days); Number of episodes/child/year with diarrhea; Number of days with vomiting.
  Recorded by the parents daily using web-based questionnaires
Fever | Up to 6 month
  Number of days with fever
  Recorded by the parents using web-based questionnaires
Antibiotic use | Up to 6 month
  Number of treatments with antibiotics during the intervention period
  Recorded weekly by the parents using web-based questionnires
Allergies | Up to 6 month
  Number of children developing allergies during the intervention period (asthma, allergic rhinitis, atopic dermatitis, food allergies); Age for diagnosis of allergies; Use of medication due to allergies.
  Recorded by the parents monthly using web-based questionnaires
Absence from day care due to illness other than infections | Up to 6 month
  Number of days the child is absent from day care due to illness, which is not due to infections.
  Recorded by the parents weekly using web-based questionnaires
Parental absence from work due to illness of the child | Up to 6 month
  Number of days a parent is absent from work due to illness of the child (infections and other illnesses, respectively)
  Recorded by the parents weekly using web-based questionnaires
Medical visits | Up to 6 month
  Number of visits to a doctor due to infections and other illnesses, respectively.
  Recorded by the parents using web-based questionnaires
Change from baseline in Thymus size | At baseline and after 6 mo (end of intervention)
  Change in thymic size during intervention period will be evaluated using ultraound

OTHER OUTCOMES:
Change from baseline in biological markers for the immune system | At baseline and after 6 mo
  Analysis of biological material investigating the effect on the immune system by biological markers .
Change from baseline in biological markers for gastro-intestinal tract | At baseline and after 6 mo
  Analysis of biological material investigating the effect on the gastrointestinal tract.
Change from baseline in Biological markers of allergy | At baseline and after 6 mo
  analysis of biological samples investigating the effect on allergy by biological markers at baseline and at 6 mo

CONTACTS AND LOCATIONS:
Locations (1):
- Section of Paediatric and International nutrition, Department of Nutrition, Exercise and Sports, Faculty of Science, University of Copenhagen, Frederiksberg, Denmark